CLINICAL TRIAL: NCT03397732
Title: Perioperative Evaluation of MMP-9-TIMP-1 System in Vascular Surgery Regarding Ischemic-reperfusion Injury
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Gábor László Woth, Principal Investigator, University of Pecs
Other Study IDs: 4330
Record Dates: First submitted 2018-01-06; First posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Ischemia Reperfusion Injury
Keywords: Matrix metalloproteinase; Tissue inhibitor of matrix metalloproteinase; Vascular surgery; Aorta stent implantation; Aorto-bifemoral bypass surgery
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aorto-bifemoral bypass: Patients scheduled for elective aorto-bifemoral bypass surgery by vascular surgeons and consented to participate in the study.
  Interventions: Procedure: aorto-bifemoral bypass and aorta stentgraft
- Aorta stentgraft: Patients scheduled for elective aorta stentgraft implantation by vascular surgeons and consented to participate in the study.
  Interventions: Procedure: aorto-bifemoral bypass and aorta stentgraft

INTERVENTIONS:
Procedure: aorto-bifemoral bypass and aorta stentgraft — Surgical implantation of aorto-bifemoral bypass or aorta stentgraft under general and/or regional anaesthesia.

SUMMARY:
The MMP-9-TIMP-1 system has been implicated in many physiological and pathophysiological conditions including vascular surgery related ischemic-reperfusion injury. Our key aims were to establish the early perioperative time courses of the aforementioned system in aorto-bifemoral bypass and aorta stentgraft implantation procedures and to find correlation between the MMP-9-TIMP-1 system and the cross-clamp time. Patients were prospectively enrolled after Ethical Committee approval. Blood samples were taken at four different time points (T1-4): T1: right before surgery, T2: 60 min after the cross-clamp release, T3: first postoperative morning, T4: third postoperative morning. Plasma was isolated from heparin anticoagulated blood samples by low speed centrifugation at 4 °C, and stored at -80 °C until analyzed in a single batch at the end of the study. MMP- 9 and TIMP-1 were determined by the quantitative sandwich enzyme-linked immunosorbent assay (ELISA) techniques according to the manufacturer instructions (R&D Systems Inc., Minneapolis, Minnesota, USA). In comparison with standard curves, the concentrations of MMP-9 and TIMP-1 in plasma were determined spectrophotometrically (Multiskan Ascent microplate photometer, Type: 354, Thermo Electron Corporation, Waltham, Massachusetts, USA) by reading the absorbance at 450 nm. Plasma concentrations of MMP-9 and TIMP-1 were expressed as ng/ml.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective procedure (aorto-bifemoral bypass or aorta stentgraft implantation) by vascular surgeons.
* Over age 18
* agree to participate

Exclusion Criteria:

* under age 18
* refuse to participate
* diagnosed malignant disease
* chronic steroid usage
* being on cytostatic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed atherosclerotic and/or aorta aneurysma generaly associated with hypertension and diabetes
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2013-06-01 (Actual)

PRIMARY OUTCOMES:
Perioperative time course of the MMP-9-TIMP-1 system | 3 days
  To establish the early perioperative time course of MMP-9-TIMP-1 system in aorto-bifemoral bypass and aorta stentgraft implantation.

SECONDARY OUTCOMES:
MMP-9-TIMP-1 system and ischemia-reperfusion injury | 3 days
  To explore relationship between MMP-9-TIMP-1 system and vascular surgery related ischemia-reperfusion injury

CONTACTS AND LOCATIONS:
Overall Officials: Diána Mühl, MD, PhD, Study Chair — University of Pécs, Dept. of Anaesthesia and Intensive Care Pécs, Baranya county, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nagy B, Szelig L, Rendeki S, Loibl C, Rezman B, Lantos J, Bogar L, Csontos C. Dynamic changes of matrix metalloproteinase 9 and tissue inhibitor of metalloproteinase 1 after burn injury. J Crit Care. 2015 Feb;30(1):162-6. doi: 10.1016/j.jcrc.2014.07.008. Epub 2014 Jul 11. PMID 25155253
- [Result] Muhl D, Nagy B, Woth G, Falusi B, Bogar L, Weber G, Lantos J. Dynamic changes of matrix metalloproteinases and their tissue inhibitors in severe sepsis. J Crit Care. 2011 Dec;26(6):550-5. doi: 10.1016/j.jcrc.2011.02.011. Epub 2011 May 6. PMID 21530151